CLINICAL TRIAL: NCT02362568
Title: Human Study of Interest on Cervical Ultrasound Exploration for Association With Criteria of Difficult Intubation in General Surgery
Brief Title: Study of Interest on Cervical Ultrasound Exploration for Association With Difficult Intubation
Acronym: TUBECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: P/2013/181
Record Dates: First submitted 2014-01-28; First posted 2015-02-13 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Intubation; Difficult
Keywords: Intubation; Difficult

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cervical ultrasound exploration (No Intervention): A cervical ultrasound exploration will be performed in all patients admitted for a planned surgery performed under general anesthesia during the stay in the postoperative room.
  Interventions: Procedure: Ultrasound cervical exploration

INTERVENTIONS:
Procedure: Ultrasound cervical exploration — The cervical ultrasound exploration will consist in the ultrasound measurement of the length between the hyoid bone and the skin and the length between the thyroid cartilage and the skin. The ultrasound cervical exploration will be performed in all patients admitted in the postoperative room after a planned surgery performed under general anesthesia.

SUMMARY:
The purpose of this study is to determine if cervical ultrasound exploration can predict difficult intubation better than main validated clinical criteria.

DETAILED DESCRIPTION:
The purpose of this study is to determine if cervical ultrasound exploration can predict difficult intubation better than main validated clinical criteria in general surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* patient consent

Exclusion Criteria:

* patient nonconsent
* age under 18
* cervical surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Sensibility, Specificity, predictive positive and negative values of US cervical measures relationship between the hyoid bone and thyroid cartilage with difficult intubation | Day 1
  The measure of the length between the hyoid bone and the skin and between the thyroid cartilage and the skin will be measured using an ultrasound cervical exploration in all patients admitted in the postoperative room after planned surgery performed under general anesthesia.

SECONDARY OUTCOMES:
Sensibility, specificity and predictive positive and negative values of validated clinical criteria for difficult intubation | Day 1
  The collect of usual clinical criteria of difficult intubation in postoperative room of patients who undergo a general anesthesia for a surgery
Mortality and morbidity of difficult intubation | Day 1
  Collect any complications (hypoxia, hypotension, tooth breakage) assigned to a difficult intubation during general anesthesia for surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Boinette Romain, MD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (2):
- France (2):
  - CHRU de Besançon, Besançon, Franche Comte
  - CHU Besancon Minjoz, Besançon